CLINICAL TRIAL: NCT04415619
Title: Evaluation of Using Buccal Pad of Fat Free Tissue Transfer With Immediate Implant Placement in the Maxillary Posterior Area
Brief Title: Using Buccal Pad of Fat Free Tissue Transfer With Immediate Implant Placement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Dina Youssef Attia, Assistant lecturer, Alexandria University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Buccal pad of fat free tissue
Record Dates: First submitted 2020-05-27; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Dental Implant
Keywords: Implant; Buccal fat pad; Immediate

STUDY DESIGN:
Intervention Model Description: A group of 10 patients will receive immediate implant placement with buccal pad of fat coverage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Intervention group (Experimental): 10 patients will have immediate implant placement with buccal pad of fat free tissue
  Interventions: Procedure: Xenograft bone substitute (Osteo-biol)

INTERVENTIONS:
Procedure: Xenograft bone substitute (Osteo-biol) — Xenograft bone substitute will be placed over the implant to cover the bone defect after extraction.
  Other Names: Implant(Superline®,DentiumCoTM); Osstell(ISQ®)

SUMMARY:
Implants placed immediately after tooth extraction usually present challenges in obtaining soft tissue coverage with high risk of bacterial invasion, wound dehiscence and subsequently adverse effect on the success rate of the implant due to lack of primary soft tissue closure over the implant.

Different surgical methods have been described to achieve primary soft tissue closure in maxillary fresh socket, each having its advantages and disadvantages, based on that, buccal pad of fat can solve this soft tissue coverage problem with minimal complications and high success rate of the placed implants.The objective of this study is to evaluate the use of buccal pad of fat tissue with immediate implant placement in the posterior maxillary area.

DETAILED DESCRIPTION:
Ten patients will be selected randomly from the outpatient clinic, Alexandria University seeking for an immediate implant placement. The sample will be selected to match the inclusion and exclusion criteria. It will be operated upon in the Oral and Maxillofacial Department, Faculty of Dentistry, Alexandria University. One stage surgery will include tooth extraction, placement of an immediate implant, bone grafting material and autologous soft tissue graft from the buccal pad of fat. Patients will be assessed clinically and radiographically to evaluate bone and soft tissue measurements.

ELIGIBILITY:
Inclusion Criteria:

* Patients age between 20-45 years with no gender predilection.
* Patients with non-restorable maxillary posterior tooth which need to be extracted (premolar -molar region).
* Patients with good oral hygiene.
* Bony defects more than 2 mm during implant placement treated by bone substitute.
* Patients fully capable to comply with the study protocol.

Exclusion Criteria:

* Patients with any systemic disease affecting bone quality as uncontrolled diabetes.
* Heavy smokers (more than 20 cigarettes per day).
* Sites with acute oral infection.
* Pregnant and lactating patients.
* Untreated periodontal disease.
* Previous chemotherapy or irradiation of the head and neck.
* Inadequate interocclusal space.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-07-01 (Estimated); Primary Completion 2020-10-13 (Estimated); Study Completion 2020-11-20 (Estimated)

PRIMARY OUTCOMES:
Evaluate postoperative pain when using the buccal pad of fat free tissue graft for primary soft tissue coverage with immediate implant placement in the posterior maxillary area. | 6 months
  Postoperative pain will be recorded by each patient after 2, 6, and 12 hours postoperatively, then daily for the first week using:
  a 10-point Visual Analogue Scale (VAS) (17) from 0 to 10 (0 no pain, to 10 severe pain).
Evaluate swelling when using the buccal pad of fat free tissue graft for primary soft tissue coverage with immediate implant placement in the posterior maxillary area. | 6 months
  Postoperative swelling will be recorded by each patient after 2, 6, and 12 hours postoperatively, then daily for the first week using a 10-point scale with 4 parameters will be used: none (no swelling), light (intraoral, localized to the treated area), moderate (extraoral swelling localized to the treated area), and severe (extraoral swelling extending beyond the treated area)
Evaluate soft tissue healing when using the buccal pad of fat free tissue graft for primary soft tissue coverage with immediate implant placement in the posterior maxillary area. | 6 months
  Evaluation of soft tissue healing
  At week 1, week4 and at 6 months:
  Presence/absence of postoperative complications will be evaluated, including:
  Bleeding, hematoma, wound dehiscence, local infection, partial flap necrosis, excessive granulation tissue or vestibular obliteration, edema, facial asymmetry and mouth opening limitation.
Evaluate implant stability when using the buccal pad of fat free tissue graft for primary soft tissue coverage with immediate implant placement in the posterior maxillary area | 6 months
  Implant stability will be measured by implant stability meter (OsstellTM), immediately postoperative and after 6 months.
Radiographic evaluation for using the buccal pad of fat free tissue graft for primary soft tissue coverage with immediate implant placement in the posterior maxillary area. | 6 months
  After 3 months then at 6 months Cone Beam CT will be requested in order to measure:
  * Bone density.
  * Amount of bone buccally and palatally to the implant.
  * Marginal bone loss.

CONTACTS AND LOCATIONS:
Overall Officials: Lobna Elwan, BSc, Principal Investigator — Alexandria University; Nagy El Prince, PhD, Study Director — Alexandria University; Ahmed O. Swedan, PhD, Study Director — Alexandria University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Penarrocha-Diago M, Alonso-Gonzalez R, Aloy-Prosper A, Penarrocha-Oltra D, Camacho F, Penarrocha-Diago M. Use of buccal fat pad to repair post-extraction peri-implant bone defects in the posterior maxilla. A preliminary prospective study. Med Oral Patol Oral Cir Bucal. 2015 Nov 1;20(6):e699-706. doi: 10.4317/medoral.20212. PMID 26241450